CLINICAL TRIAL: NCT02112071
Title: Diabetic Kidney Disease: Influence of Exercise Therapy on Physical and Vascular Function.
Acronym: DKD-EXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0905M66282; K23DK082638-04 (NIH); 22275 (Other: University of Minnesota)
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Focus Type 2 Diabetes Related Chronic Kidney Disease
Keywords: Exercise; Diabetic kidney disease; vascular function; physical function
MeSH Terms: conditions — Motor Activity; Diabetic Nephropathies | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): blended supervised-hombased exercise training 3-4 times/week for 12 weeks
  Interventions: Behavioral: Exercise
- control (No Intervention): control group asked to continue usual activities

INTERVENTIONS:
Behavioral: Exercise — Blended supervised-home based walking program 3-4 times per week for at least 30 minutes.
  Arms: Exercise

SUMMARY:
The general objective is to investigate the effect of a 12 week walking exercise program on vascular endothelial function, arterial stiffness/compliance, and vascular health biomarkers in men and women with pre-dialysis type 2 diabetic kidney disease (DKD).

ELIGIBILITY:
Inclusion Criteria:

* • An individual must be >18 years of age

Have diagnosed type 2 diabetic mellitus by one of the following criteria:

o Treated with diet, diet plus oral hypoglycemic agents (for at least one year), or insulin preceded by treatment with oral agents (for at least one year).

If treated with insulin, the onset of diabetes must have occurred after age of 40 and the body mass index must be >25kg/m2 at the time of diagnosis.

Diagnosed kidney attributed to diabetes by one of the following criteria:3

* Macroalbuminuria (ACR >300mg/g, or)
* Microalbuminuria (ACR between 30-300 mg/g) or in the presence of diabetic retinopathy (although is recognized that about 1/3 of type 2 diabetics do not have retinopathy by fundoscopic exam).
* An elevated ACR should have been confirmed in the absence of urinary tract infections with 2 additional first-void specimens collected over 3-6 months.
* At least 2 of 3 samples should fall within the range of micro or macroalbuminuria.

  * An estimated Glomerular filtration rate (GFR) of between 90 ml/min and 30 ml/min measured by (GFR (mL/min/1.73 m2) = 186 x (Scr)-1.154 x (Age)-0.203 x (0.742 if female) x (1.210 if African-American) (conventional units).
  * Individuals must be able to provide informed consent
  * Perform walking exercise testing on a treadmill
  * Be able to participate in a 12-week supervised exercise program.

Exclusion Criteria:

* • Patients are currently exercising

  * Requiring dialysis
  * Have an Hematocrit <30%
  * Uncontrolled hypertension (>200/100mmHg)
  * Peripheral vascular disease.
  * An inability to understand English or give consent. Other exclusion criteria are: any contraindications to exercise testing or training as indicated by the American College of Sports Medicine guidelines such as: Unstable coronary heart disease and symptomatic heart failure, exercise capacity limited by health problems such as angina, severe arthritis, or extreme dyspnea on exertion, progressive neuromuscular disease, pulmonary disease., or having undergone a coronary revascularization within the past 6 months prior to enrollment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-10; Primary Completion 2012-11 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
endothelial function measured by brachial artery flow mediated vasodilation | at week 0 and at week 12
  Endothelium-mediated change in in vascular tone

SECONDARY OUTCOMES:
arterial stiffness measured by pulse wave velocity | at week 0 and at week 12
Circulating markers of vascular health | at week 0 and at week 12
  C-reactive protein, isoprostane F2, Asymmetric dimethylarginine
aerobic capacity | at week 0 and at week 12
  Peak oxygen consumption
blood pressure | at week 0 and at week 12
24-hour albuminuria | at week 0 and at week 12
  assessed in 30 participants measured in milligram per gram creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Ulf G Bronas, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States